CLINICAL TRIAL: NCT00979316
Title: Randomized, Double-Blinded, Placebo-Controlled, Open Label Positive- Controlled, Four-Way Crossover Study of the Electrocardiographic Effects of BMS-708163 in Healthy Subjects
Brief Title: Effect on the Electrocardiographic QT Interval Corrected for Heart Rate (QTc) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: CN156-020
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-708163 (800 mg) (Experimental)
  Interventions: Drug: BMS-708163
- BMS-708163 (200 mg) (Experimental)
  Interventions: Drug: BMS-708163
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: BMS-708163 — Oral Solution, Oral, 800 mg, Once on Day 1, approximately 14 days
  Arms: BMS-708163 (800 mg)
Drug: BMS-708163 — Oral Solution, Oral, 200 mg, Once on Day 1, approximately 14 days
  Arms: BMS-708163 (200 mg)
Drug: Placebo — Oral Solution, Oral, 0 mg, Once on Day 1, approximately 14 days
  Arms: Placebo
Drug: Moxifloxacin — Tablets, Oral, 400 mg, Once on Day 1, approximately 14 days
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to determine the effect of BMS-708163 on the QTc interval (QT interval corrected for heart rate).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive.
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) and men, ages 18 to 55
* Healthy subjects

Exclusion Criteria:

* History of cardiac arrhythmias or palpitations associated with presyncope or syncope, or history of unexplained syncope
* Sexually active fertile men not using effective birth control (double barrier) if their partners are WOCBP
* Women who are pregnant or breastfeeding
* History of allergy or intolerance to moxifloxacin or any member of the quinolone class of antimicrobial agents
* History of hypokalemia, history or family history of prolonged QT interval, or family history of sudden cardiac death at a young age
* Any clinically significant ECG abnormality
* History of seizure disorders
* History of drowning survival

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Effect on the electrocardiographic QT interval corrected for heart rate (QTc) in healthy subjects | Serial triplicate ECGs at -60, -40 and -20 minutes prior to dosing: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 16 and 22.5 hours after dosing on Day 1 in each period

SECONDARY OUTCOMES:
To assess the effects of BMS-708163 on other ECG endpoints (heart rate [HR], QRS and PR intervals), and changes in waveform morphology | At -60, -40 and -20 minutes prior to dosing; at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 16 and 22.5 hours after dosing on Day 1 in each period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services (Us), Inc, Tempe, Arizona, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx